CLINICAL TRIAL: NCT06431061
Title: Clinical Evaluation of Proclear Toric and Biofinity Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-158
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (omafilcon B) (Experimental): All participants will wear lens A for 15 minutes (Period 1).
  Interventions: Device: Lens A (omafilcon B)
- Lens B (comfilcon A) (Experimental): All participants will wear lens B for 15 minutes (Period 2).
  Interventions: Device: Lens B (comfilcon A)

INTERVENTIONS:
Device: Lens A (omafilcon B) — 15 minutes of daily wear.
  Arms: Lens A (omafilcon B)
Device: Lens B (comfilcon A) — 15 minutes of daily wear.
  Arms: Lens B (comfilcon A)

SUMMARY:
The aim of this study is to compare the short-term clinical performance of two Toric contact lenses.

DETAILED DESCRIPTION:
The aim of the study is to evaluate and compare the performance of two soft toric contact lenses in existing soft toric lens wearers in a short term (15 minutes wear) study.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 17 years of age and has full legal capacity to volunteer.
2. Have understood and signed an information consent letter.
3. Are willing and able to follow instructions and maintain the appointment schedule.
4. Are an adapted soft toric contact lens wearer.
5. Do not habitually wear either of the two study lens types.
6. Have a vertex-corrected contact lens prescription with a spherical component of +4.00D to -9.00D in combination with astigmatism of no less than -0.75D and no more than -2.25D in each eye.
7. Can achieve best corrected distance visual acuity of +0.10 logMAR (subjective refraction) or better in each eye.
8. Can be fitted with and achieve a distance visual acuity of +0.18 logMAR or better in each eye with the study contact lenses.

Exclusion Criteria:

1. Are participating in any concurrent clinical or research study.
2. Have any known active ocular disease and/or infection or slit lamp findings that would contraindicate contact lens use.
3. Have a systemic condition that in the opinion of the investigator may affect a study outcome variable.
4. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable.
5. Have known sensitivity to the diagnostic pharmaceuticals to be used in the study.
6. Have a history of not achieving comfortable CL use (5 days per week; > 8 hours/day)
7. Are an employee of the Centre for Ocular Research & Education directly involved in the study (i.e. on the delegation log).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — Centre for Ocular Research and Education
Locations (1):
- University of Waterloo, Waterloo, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-eight Participants were screened. One Participant was not eligible due to screening failure.
  All the participants who were eligible in the study were included in the analysis. (n=37)
Groups:
- Lens A (Omafilcon B): All participants wore lens A for 15 minutes (Period 1).
  Lens A (omafilcon B): 15 minutes of daily wear.
- Lens B (Comfilcon A): All participants wore lens B for 15 minutes (Period 2).
  Lens B (comfilcon A): 15 minutes of daily wear.
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A (Omafilcon B) | Lens B (Comfilcon A)
Started | 37 | 0 (All participants received Lens A in Period 1.)
Completed | 37 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A (Omafilcon B) | Lens B (Comfilcon A)
Started | 0 (All participants received Lens B in Period 2.) | 37
Completed | 0 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Fit Acceptance
Description: Overall fit acceptance will be measured on scale of (0-4) where (0=Should not be worn and 4=Perfect)
Time Frame: After 15 minutes of continuous wear
Population: All the participants who were eligible in the study were included in the analysis. (n=37)
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Lens A (Omafilcon B) | Lens B (Comfilcon A)
Number analyzed (Participants) | 37 | 37
Units on Scale | 3.5 (0.7) | 3.8 (0.4)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 23 weeks
Arm/Group | Lens A (Omafilcon B) | Lens B (Comfilcon A)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT06431061/Prot_SAP_000.pdf